CLINICAL TRIAL: NCT04431284
Title: Impact of COVID-19 Lockdown on Severely Obese Patients With or Without Binge Eating Behaviors
Brief Title: Impact of COVID-19 Lockdown on Obesity and Eating Behaviors
Acronym: CIO
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0516; 2020-A01616-33 (Other: ID-RCB)
Record Dates: First submitted 2020-06-10; First posted 2020-06-16 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Feeding and Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obese patients with binge eating disorders: Severely obese patients (with or without binge eating disorders, Binge Eating Sclae >= 16) who have been hospitalized for obesity assessment before the start of the lockdown in the Endocrinology department of the Lyon Hospital
  Interventions: Other: Questionnaires
- Obese patients without binge eating disorders: Severely obese patients (with or without binge eating disorders, Binge Eating Sclae >= 16) who have been hospitalized for obesity assessment before the start of the lockdown in the Endocrinology department of the Lyon Hospital
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — The two groups (23 patients per group) will be contacted by phone or e-mail to participate to the CIO study. Once their agreement received, each patient will be asked to complete the same set of online questionnaires : weight, HAD (Hospital Anxiety and Depression scale), BES (Binge Eating Scale), YFAS (Yale Food Addiction Scale), DEBQ (Dutch Eating Behavior Questionnaire), IPAQ (International physical activity questionnaire), COVID 19 questionnaire Penn State, items from the Do-It questionnaire, general questions on the lifestyle during the lockdown (custom questionnaire), COVID stress evaluation (custom questionnaire)

SUMMARY:
COVID-19 lockdown presents particular challenges for people living with obesity. Indeed during this period, the lifestyle was deeply modified: diet, activity, and sleep behaviours, home office, take care of child, social distancing... All of these modifications may have led to stress and anxiety. It has been previously demonstrated that high perceived stress levels are correlated with high preference for sweet and fat foods . In this context caution would be exercised in obese patients especially those with binge eating disorders. Indeed binge eating disorder is characterized by compulsive overeating or consuming abnormal amounts of food while feeling unable to stop and a loss of control. And one key trigger of binge eating disorder is stress and anxiety. Thus, patients with binge eating disorders may have been more sensitive to the impact of lockdown and thus urgently would require appropriated care management.

The main objective is to compare the eating behaviour between obese patients with or without binge eating disorders. The second objective is to compare the weight evolution between the two groups before and after the lockdown.

To reach these objectives, the scientific team of the CIO project proposes to contact by phone and e-mail obese patients (with or without binge eating disorders) who have been hospitalized for their obesity disease before the start of the lockdown in the Endocrinology department of the Lyon Hospital. The patients will be asked to fill in several questionnaires (using an online tool) allowing to evaluate their mood, anxiety, eating behaviour, binge eating disorders… during the lockdown. The results of these questionnaires will be compared to those collected during their hospitalisation before the lockdown.

The hypothesis is that participants suffering from binge eating disorder will have more sever eating behaviour perturbations as higher level of stress, anxiety, depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* severely obese patients

Exclusion Criteria:

* patients do not experiment the full lockdown period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients with or without binge eating disorders
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
Comparison of the BMI (kg/m²) evolution between the two groups | Day 21
Score comparison of the Dutch Eating Behavior Questionnaire | Day 21

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel DISSE, MD, Principal Investigator — Centre Intégré de l'obésité de Lyon / HCL; Martine LAVILLE, MD, Principal Investigator — Centre Intégré de l'obésité de Lyon / HCL
Locations (1):
- Centre Intégré de l'obésité de Lyon / HCL, Pierre-Bénite, France

REFERENCES:
- [Background] Torres SJ, Nowson CA. Relationship between stress, eating behavior, and obesity. Nutrition. 2007 Nov-Dec;23(11-12):887-94. doi: 10.1016/j.nut.2007.08.008. Epub 2007 Sep 17. PMID 17869482